CLINICAL TRIAL: NCT04880317
Title: Validation of Quantitative Myocardial Tissue Characterization Through Contrast-enhanced Non-gated CT Versus CMR: The VALETUDO-CT Study
Brief Title: Validation of Quantitative Myocardial Tissue Characterization Through Non-gated CT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI ceased activity
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco Sardanelli, Head of Radiology, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VALETUDO
Record Dates: First submitted 2021-05-02; First posted 2021-05-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Disease; Covid19; Cardiotoxicity; Extracellular Space Alteration
Keywords: Tomography X-Ray Computed; Magnetic Resonance Imaging; Cardiotoxicity; Extracellular Space
MeSH Terms: conditions — Heart Diseases; COVID-19; Cardiotoxicity | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance; Diagnostic Test: Additional CT acquisition; Diagnostic Test: Blood tests

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance — All enrolled patients will undergo a contrast-enhanced CMR examination for the assessment of extracellular volume
Diagnostic Test: Additional CT acquisition — All enrolled patients will undergo an additional CT scan at 5 minutes post-contrast injection to evaluate myocardial relative enhancement
Diagnostic Test: Blood tests — Patients will undergo blood tests to review hematocrit, Sars-CoV-2 antibody status and cardiac fibrosis biomarkers

SUMMARY:
The main aim is to validate non-gated 5-min computed tomography myocardial relative enhancement (CT-MRE), which can be readily estimated via contrast-enhanced non-gated chest CT, as a tool for estimating myocardial extracellular volume (ECV) using cardiac magnetic resonance (CMR)-derived ECV as a reference standard in a consecutive series of patients scheduled for cardiac CT.

A secondary explorative aim is to evaluate the presence and extent of possible myocardial alterations in those patients enrolled in the VALETUDO study who have been infected with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

DETAILED DESCRIPTION:
Patients scheduled to undergo contrast-enhanced cardiac CT and meeting inclusion criteria will be proposed enrolment in the study, and as such they will be informed on the study aims and design and will be invited to sign a specific informed consent. All potential enrollees will be invited to undergo an additional CT acquisition as part of their cardiac CT examination, to estimate CT-MRE, blood tests, and a contrast-enhanced CMR scan. All those meeting exclusion criteria (contraindications to CMR, previous allergic reactions to gadolinium-based contrast agents, pregnancy, severe obesity, claustrophobia) will be consequently excluded from the study. Patients with a previous diagnosis of COVID-19 will not be excluded if they are declared negative according to the procedure provided for by the regulations in force.

For all those eventually included to participate in the study, the CT examination will include the addition of a non-gated 5-min delayed acquisition, allowing the assessment of CT-MRE. All enrolled patients will then undergo blood tests including the assessment of haematocrit for the calculation of ECV and CT-MRE, and serological testing for COVID-19 antibodies. An additional blood sample (for a total of 30 ml of venous blood) will be tested for myocardial fibrosis biomarkers (Troponin, Osteopontin, ST, and Osteocalcin), and the remaining samples will be long-term bio-banked pending patients' approval.

All enrolled patients will then undergo a CMR examination within 10 days of the cardiac CT scan, including the intravenous administration of a macrocyclic gadolinium-based contrast agent, including cine sequences for myocardial function and strain assessment, and native- and contrast-enhanced T1 mapping for myocardial ECV calculation.

Myocardial CT-MRE and CMR-derived ECV calculation will be conducted according to methods previously described by the two centres. All CT and CMR exams will be anonymized, and segmentation for such purposes will be performed by readers with extensive experience in cardiovascular CT and CMR. Additionally, myocardial strain will be calculated from CMR cine sequences, through dedicated software.

Taking into consideration the known correlation between CT- and CMR-derived ECV and given the correlation between CT-MRE and CT-derived ECV noted in a previous study from our group, we would expect the coefficient of the correlation between CT-MRE and CMR-derived ECV not to be lower than 0.3. On these grounds, aiming for an α error of 0.05 and a statistical power (1 - β) of 0.90, we would require a sample size of 113 patients for our principal aim. Considering a potential maximum dropout rate around 40% (mostly due to the refusal to undergo CMR on a subsequent date from cardiac CT), we aim to enrol 188 patients for our study.

Normality will be evaluated using Shapiro-Wilk test. In case of normal distribution, t-tests will be used to assess differences between groups, and Pearson's r will be used for correlations. In case of non-normal distributions, Mann-Whitney and Wilcoxon tests will be used to assess differences, and Spearman's ρ for correlations. P-values ≤0.05 will be considered as indicative of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for contrast-enhanced cardiac CT
* Age 18 to 80 years

Exclusion Criteria:

* Absolute contraindications to CMR
* Implantable cardioverter defibrillators and ferromagnetic thoracic devices which may cause artifacts at magnetic resonance imaging
* Previous allergic reactions to gadolinium-based contrast agents
* Pregnancy
* Severe obesity
* Severe claustrophobia
* Too low image quality to perform post-processing analyses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Validation of CT-MRE as a surrogate of CMR-ECV | 3 months
  CT-MRE will be calculated as (1-hematocrit) multiplied by the ratio of the differences in image density between post- and pre-contrast images in the myocardium and blood pool. Thus, CT-MRE will be represented by a percentage value. It will be calculated by placing regions of interest on the appropriate CT images.

SECONDARY OUTCOMES:
Assessment of correlations between CMR-derived myocardial strain, CMR-ECV and CT-MRE | 3 months
  Myocardial strain will be calculated via feature tracking algorithms, segmenting the endocardium and epicardium on cine images. As strain represents the ratio between the difference in displacement of the myocardial wall and its original position, it will be represented by a percentage. Strain will be measured in its longitudinal, radial and circumferential components.
Role of ECV as a biomarker of chronic cardiac damage following SARS-CoV-2 infection | 3 months
  ECV will be calculated as the product between (1-hematocrit) and the ratio of the differences in image intensity between pre- and post-contrast T1 maps in the myocardium and blood pool. Data for this calculation will be derived by placing regions of interest in the appropriate MRI T1 maps. ECV is thus represented by a percentual value

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided